CLINICAL TRIAL: NCT07252583
Title: Relationships Between Sexuality and Mental Health in Older People
Acronym: PASS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RNI 2025 LAHAYE; 2025-A01231-48 (Other: ANSM)
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Old Age
Keywords: sexuality
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all patients are enrolled prospectively. No comparator (Experimental): questionnaires arm
  Interventions: Other: questionnaires of quality of life

INTERVENTIONS:
Other: questionnaires of quality of life — patient self-administered questionnaires

SUMMARY:
The prevalence of sexual activity decreases with age, particularly among individuals over 60 years old. Although physical dysfunctions, such as erectile disorders, play a role, the decline in sexuality is also linked to cultural and social factors, such as stereotypes and the loss of a partner. Sexuality in adulthood impacts both mental and physical health, contributing to better quality of life and reduced risks of cardiovascular disease and cancer. Maintaining a fulfilling sexual life among older adults is a public health issue that remains underexplored, particularly regarding its relationship with mental health.

Primary objective To explore the association between sexuality and mental health in community-dwelling older adults.

Secondary objectives To study the relationships between the different dimensions of the questionnaires (ISS, QLQC30, HAD) To examine the association between sexuality and psychotropic drug use To compare sexuality and mental health among older adults belonging to senior associations and those living in independent residences

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participant aged ≥ 60 years (male or female)

Exclusion Criteria:

* Inability to understand or communicate in French
* Major neurocognitive disorders
* Refusal to participate in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety Depression Scale HAD Quality of Life Questionary QLQC30 Index of Sexual Satisfaction ISS | Day 1 Inclusion
  Analysis will focus on questionnaire scores

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Gabriel Montpied, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Undecided